CLINICAL TRIAL: NCT03392155
Title: The Effectiveness of a Performance and Nutrition Program for Athletes in Adaptive Sports
Brief Title: Performance and Nutrition Program for Athletes in Adaptive Sports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Meegan G. Van Straaten, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-005392
Record Dates: First submitted 2017-12-26; First posted 2018-01-05 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injuries; Physical Disability
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training & Nutrition (Experimental): Participants receive performance training twice a week for 12 weeks and group and individual nutritional counseling during the 12 weeks.
  Interventions: Behavioral: Training & Nutrition

INTERVENTIONS:
Behavioral: Training & Nutrition — Exercise at moderate to high intensities and diet education/counseling

SUMMARY:
Researchers are trying to evaluate and recommend sustainable and effective health and wellness programs for people with spinal cord injury (SCI) and other physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

Group1 (Group with spinal cord injury):

* Participants with traumatic or non-traumatic spinal cord injury
* Able to perform progressive exercise program
* Willingness to participate in study

Group 2 (Able-bodied group):

* Functional upper extremity range of motion
* Able to perform progressive exercise program
* Willingness to participate in study

Group3 (Other physical disability group):

* Participants with a physical disability other than spinal cord injury
* Able to perform progressive exercise program
* Willingness to participate in study

Exclusion Criteria:

All groups:

• Any documented or reported health condition that would be contraindicated to a progressive exercise program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in The World Health Organization Quality of Life Score (WHOQOL-BREF) | Baseline (during week 1-2 of study), After intervention (week 16), 12 weeks after completion of study (week 28)
  The World Health Organization (WHOQOL-BREF) is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health. Each domain's mean score can range between 4 and 20 and a higher score indicates a higher quality of life.

SECONDARY OUTCOMES:
Change in exercise self-efficacy score (for participants not living with spinal cord injury) | Baseline (during week 1-2 of study), After intervention (week 16), 12 weeks after completion of study (week 28)
  The Barriers Specific Self-Efficacy Scale is a self-reported survey and was designed to measure subjects' perceived capabilities to exercise even if faced with barriers to exercise. Scores can range from zero to 100 with higher numbers indicating better confidence that the subject has the capability to exercise.
Change in exercise self-efficacy score (for participants living with spinal cord injury) | Baseline (during week 1-2 of study), After intervention (week 16), 12 weeks after completion of study (week 28)
  The Spinal Cord Injury Exercise Self-Efficacy Scale (ESES) is a self-reported survey and includes 10 questions and a maximum score of 40 with higher scores indicating more confidence to exercise.
Change in self-reported un-weighed food records | Baseline (during week 1-2 of study), After intervention (week 16), 12 weeks after completion of study (week 28)
  Self-reported un-weighed food records are collected by participant interview with a registered dietician and also with digital photography of full food plates and left-overs. Improvement in dietary intake is indicated from a "yes" or "no" of whether study participants have met individual goals that are determined during baseline session with dietician.

CONTACTS AND LOCATIONS:
Overall Officials: Meegan G Van Straaten, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials